CLINICAL TRIAL: NCT00229476
Title: Study of Medication and Placebo Response in Major Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Eli Lilly and Company (Industry); Pfizer (Industry); Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 03-08-033; H6U-US-X002; 04012549
Record Dates: First submitted 2005-09-28; First posted 2005-09-29 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Depressive Disorder, Major
Keywords: Depression; EEG; QEEG; cordance; Zoloft; sertraline; placebo; electroencephalogram; brain; antidepressants
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Sertraline

INTERVENTIONS:
Drug: sertraline (Zoloft)

SUMMARY:
The primary purpose of the research study is to use recordings of brain electrical activity (through electroencephalogram, or EEG) and symptom measurements to determine whether patients are likely to show a response to medication or placebo treatment during a treatment trial for depression.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Unipolar Major Depression

Exclusion Criteria:

* Substance Abuse, Psychotic Disorder, History of Severe Head Trauma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-12; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
depressive symptoms

SECONDARY OUTCOMES:
brain electrical activity (EEG)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew F. Leuchter, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Neuropsychiatric Institute & Hospital, Los Angeles, California, United States

REFERENCES:
- [Background] Leuchter AF, Cook IA, Witte EA, Morgan M, Abrams M. Changes in brain function of depressed subjects during treatment with placebo. Am J Psychiatry. 2002 Jan;159(1):122-9. doi: 10.1176/appi.ajp.159.1.122. PMID 11772700
- [Background] Cook IA, Leuchter AF, Morgan M, Witte E, Stubbeman WF, Abrams M, Rosenberg S, Uijtdehaage SH. Early changes in prefrontal activity characterize clinical responders to antidepressants. Neuropsychopharmacology. 2002 Jul;27(1):120-31. doi: 10.1016/S0893-133X(02)00294-4. PMID 12062912
- [Background] Leuchter AF, Morgan M, Cook IA, Dunkin J, Abrams M, Witte E. Pretreatment neurophysiological and clinical characteristics of placebo responders in treatment trials for major depression. Psychopharmacology (Berl). 2004 Dec;177(1-2):15-22. doi: 10.1007/s00213-004-1919-2. Epub 2004 Jul 14. PMID 15252704
- See also: Depression Research at UCLA - Click here for more information about this study: Study of Medication and Placebo Response in Major Depression — http://www.DepressionResearch.com/